CLINICAL TRIAL: NCT03496506
Title: A Single-center, Open-label, Two-treatment, One-sequence, Cross-over Study to Investigate the Effect of Clopidogrel on the Pharmacokinetics of Selexipag and Its Active Metabolite, ACT-333679, in Healthy Male Subjects
Brief Title: A Clinical Study to Assess the Effect of Clopidogrel on the Pharmacokinetics of Selexipag and Its Active Metabolite in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-065-117
Record Dates: First submitted 2018-04-06; First posted 2018-04-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects
Keywords: selexipag; clopidogrel
MeSH Terms: interventions — selexipag; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Open-label, two-treatment, one-sequence, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential treatment arm (Experimental): Subjects receive 1 tablet of selexipag twice daily from Day 1 to Day 9 and 1 tablet in the morning of Day 10. In the morning of Day 4 and 1 hour before the administration of selexipag, they receive 4 tablets of clopidogrel. Then from Day 5 to Day 10, 1 hour before the morning administration of selexipag, they receive 1 tablet of clopidogrel .
  Interventions: Drug: Selexipag; Drug: Clopidogrel

INTERVENTIONS:
Drug: Selexipag — Each film-coated tablet contains 200 microgram (mcg) of selexipag (oral use)
  Other Names: ACT-293987
Drug: Clopidogrel — Each film-coated tablet containing 75 mg of clopidogrel (oral use)

SUMMARY:
The purpose of this study is to evaluate the effect of clopidogrel on the pharmacokinetics of selexipag and its active metabolite (ACT-333679) in healthy male adults (by determining the blood concentrations of selexipag and its metabolite). Also, the safety of selexipag when administered alone or with clopidogrel will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Healty male subjects aged between 18 and 45 years (inclusive) at screening.
* Body mass index from 18.0 to 28.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 45-90 bpm (inclusive).

Exclusion Criteria:

* Any contraindication included in the SmPC of selexipag or clopidogrel treatment.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatments.
* History or clinical evidence of any disorder of hemostasis, hemorrhagic diathesis, nose or gingival bleeding, hemophilia, thrombotic thrombocytopenic purpura, presence of any lesions with a propensity to bleed (particularly gastrointestinal and intraocular), history of bleeding complications after surgical procedures such as tooth extraction
* Previous history of stroke, fainting, collapse, syncope, orthostatic hypotension,vasovagal reactions, head injury.
* Excessive caffeine consumption
* Nicotine consumption within 3 months prior to screening, and inability to refrain from nicotine consumption during the course of the study
* Previous treatment with any prescribed medications (including vaccines) or over the counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks prior to first selexipag administration.
* Subjects with rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile of selexipag and ACT-333679 during a dose interval (AUC-tau) | Blood samples at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dose on Day 3, Day 4 and Day 10
  AUC-tau for selexipag and ACT-333679 is calculated on the basis of the actual blood sampling time points drawn during the 12-hour interval after the morning administration of selexipag administered either alone (Day 3) or concomitantly with clopidogrel (Day 4 and Day 10)
Maximal plasma concentration of selexipag and ACT-333679 (Cmax) | Blood samples at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dose on Day 3, Day 4 and Day 10
  Cmax is directly derived from the individual plasma concentration-time curves for selexipag and ACT-333679, following administration of selexipag alone (Day 3) or concomitantly with clopidogrel (Day 4 and Day 10)

SECONDARY OUTCOMES:
Trough plasma concentration of selexipag and ACT-333679 (Ctrough) | Blood samples from Day 1 to Day 9 before the morning and evening administrations of selexipag and on Day 10 before the morning administration of selexipag
  Ctrough is the concentration of selexipag and ACT-333679 directly measured in the blood samples collected prior to the morning and evening administrations of selexipag
Time to reach Cmax (tmax) | Blood samples at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dose on Day 3, Day 4 and Day 10
  tmax is the time to reach the maximal plasma concentration of selexipag and ACT-333679 and it is directly derived from the individual plasma concentration-time curves for selexipag and ACT-333679, following administration of selexipag alone (Day 3) or concomitantly with clopidogrel (Day 4 and Day 10)
Number of participants with any treatment-emergent adverse events (TEAEs) including serious adverse events | From the first selexipag administration on Day 1 up to Day 18 (about 1 week after the last administration of selexipag)
  A treatment-emergent adverse event is any adverse event temporally associated with the use of a study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Bruderer, Study Director — Actelion
Locations (1):
- Clinical Pharmacology Unit (CPU), Merksem, Belgium

REFERENCES:
- [Derived] Axelsen LN, Poggesi I, Rasschaert F, Perez Ruixo JJ, Bruderer S. Clopidogrel, a CYP2C8 inhibitor, causes a clinically relevant increase in the systemic exposure to the active metabolite of selexipag in healthy subjects. Br J Clin Pharmacol. 2021 Jan;87(1):119-128. doi: 10.1111/bcp.14365. Epub 2020 Jun 5. PMID 32415684